CLINICAL TRIAL: NCT07260708
Title: A Phase I Clinical Study to Evaluate The Safety and Pharmacokinetics of TQB2922 Injection (Subcutaneous Injection) in Patients With Advanced Cancers
Brief Title: Clinical Trial of TQB2922 Injection (Subcutaneous Injection) in Patients With Advanced Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Chia Tai Tianqing Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2922-I-02
Record Dates: First submitted 2025-11-20; First posted 2025-12-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-09

CONDITIONS: Advanced Cancers
MeSH Terms: interventions — Injections, Subcutaneous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2922 injection (subcutaneous injection) (Experimental): TQB2922 injection (Subcutaneous Injection), 28 days as a treatment cycle
  Interventions: Drug: TQB2922 injection (subcutaneous injection)

INTERVENTIONS:
Drug: TQB2922 injection (subcutaneous injection) — TQB2922 is a bispecific antibody against Epidermal Growth Factor Receptor (EGFR)/c-Met.

SUMMARY:
This is a Phase I clinical study aimed at evaluating the safety and pharmacokinetics of TQB2922 subcutaneous injection in patients with advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily joined this study, signed the informed consent form, and had good compliance；
* 18-75 yeas old；
* Eastern Cooperative Oncology Group Performance Status (ECOG) score: 0-1;
* Expected survival of more than 12 weeks；
* Histologically or cytologically diagnosed with advanced non-squamous non-small cell lung cancer
* Subjects in the monotherapy introduction stage need to have received standard treatment or lack effective treatment.
* There must be at least one measurable lesion within the radiotherapy area that can be clearly classified as progressive according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST1.1) criteria.
* Major organs are functioning well；
* Female and male subjects of childbearing potential should agree to practice contraception for the duration of the study and for 6 months after the end of the study.

Exclusion Criteria:

* Current concomitant presence of other malignancies within 5 years prior to the first dose；
* At the time of initiating the study of treatment, the adverse reactions caused by previous anti-tumor treatments failed to recover to a CTCAE 5.0 score of grade 1 or below.
* Patients who had received major surgical treatment within 4 weeks prior to the first study, had obvious traumatic injuries, or were expected to undergo major surgery during the study treatment period, or had long-term unhealed wounds or fractures.
* Hyperactive or venous thrombosis events occurred within 6 months before the first administration;
* Major cardiovascular diseases;
* Active hepatitis
* Those with a history of psychotropic drug abuse who are unable to quit or have mental disorders.
* There was an active infection (≥ Common Terminology Criteria for Adverse Events version 5.0 (CTCAE5.0) score of grade 2) within 2 weeks before the first administration;
* Patients with renal failure requiring hemodialysis or peritoneal dialysis;
* Patients who have a history of immune deficiency.
* Patients who have epilepsy and need treatment;
* Evidence of a previous history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid treatment, or any clinically active interstitial lung disease.
* Those who have participated in and used other anti-tumor clinical trial drugs within 4 weeks before the first treatment.
* Pregnant or lactating women.
* There is any serious or uncontrolled systemic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Time to Peak Concentration | Cycle 1 Day 1:predose, 2, 6, 10, 24, 48, 72 hours after infusion, Cycle 1 Day 8, 15, 22:predose; Cycle 2 Day1: predose, 2, 6 h, 10, 24, 48, 72, 168 hours after infusion; Cycle 2 Day 15;Day 1 on Cycle 4, Cycle 6,Cycle 8: predose (each cycle is 28 days)
  Time to Peak Concentration
Peak concentration | Cycle 1 Day 1:predose, 2, 6, 10, 24, 48, 72 hours after infusion, Cycle 1 Day 8, 15, 22:predose; Cycle 2 Day1: predose, 2, 6 h, 10, 24, 48, 72, 168 hours after infusion; Cycle 2 Day 15;Day 1 on Cycle 4, Cycle 6,Cycle 8: predose (each cycle is 28 days)
  Maximum plasma drug concentration
half-life (T1/2) | Cycle 1 Day 1:predose, 2, 6, 10, 24, 48, 72 hours after infusion, Cycle 1 Day 8, 15, 22:predose; Cycle 2 Day1: predose, 2, 6 h, 10, 24, 48, 72, 168 hours after infusion; Cycle 2 Day 15;Day 1 on Cycle 4, Cycle 6,Cycle 8: predose (each cycle is 28 days)
  Terminal half-life (T1/2)
The area under the curve (AUC0-∞） | Cycle 1 Day 1:predose, 2, 6, 10, 24, 48, 72 hours after infusion, Cycle 1 Day 8, 15, 22:predose; Cycle 2 Day1: predose, 2, 6 h, 10, 24, 48, 72, 168 hours after infusion; Cycle 2 Day 15;Day 1 on Cycle 4, Cycle 6,Cycle 8: predose (each cycle is 28 days)
  The area under the plasma concentration-time curve extrapolated from the first administration to infinity
The area under the curve (AUC0-t) | Cycle 1 Day 1:predose, 2, 6, 10, 24, 48, 72 hours after infusion, Cycle 1 Day 8, 15, 22:predose; Cycle 2 Day1: predose, 2, 6 h, 10, 24, 48, 72, 168 hours after infusion; Cycle 2 Day 15;Day 1 on Cycle 4, Cycle 6,Cycle 8: predose (each cycle is 28 days)
  The area under the plasma concentration-time curve from the time of the first administration to the last quantifiable concentration time point.
Elimination Rate | Cycle 1 Day 1:predose, 2, 6, 10, 24, 48, 72 hours after infusion, Cycle 1 Day 8, 15, 22:predose; Cycle 2 Day1: predose, 2, 6 h, 10, 24, 48, 72, 168 hours after infusion; Cycle 2 Day 15;Day 1 on Cycle 4, Cycle 6,Cycle 8: predose (each cycle is 28 days)
  Reflects the rate at which a drug disappears from the bloodstream
Apparent Oral Clearance | Cycle 1 Day 1:predose, 2, 6, 10, 24, 48, 72 hours after infusion, Cycle 1 Day 8, 15, 22:predose; Cycle 2 Day1: predose, 2, 6 h, 10, 24, 48, 72, 168 hours after infusion; Cycle 2 Day 15;Day 1 on Cycle 4, Cycle 6,Cycle 8: predose (each cycle is 28 days)
  The mixed effect reflecting the drug's clearance ability and absorption degree.
Apparent Volume of Distribution | Cycle 1 Day 1:predose, 2, 6, 10, 24, 48, 72 hours after infusion, Cycle 1 Day 8, 15, 22:predose; Cycle 2 Day1: predose, 2, 6 h, 10, 24, 48, 72, 168 hours after infusion; Cycle 2 Day 15;Day 1 on Cycle 4, Cycle 6,Cycle 8: predose (each cycle is 28 days)
  The mixed effect reflecting the degree of drug distribution and absorption.
Trough Concentration | Cycle 1 Day 1:predose, 2, 6, 10, 24, 48, 72 hours after infusion, Cycle 1 Day 8, 15, 22:predose; Cycle 2 Day1: predose, 2, 6 h, 10, 24, 48, 72, 168 hours after infusion; Cycle 2 Day 15;Day 1 on Cycle 4, Cycle 6,Cycle 8: predose (each cycle is 28 days)
  The blood drug concentration at the moment before the next administration.
Accumulation Ratio | Cycle 1 Day 1:predose, 2, 6, 10, 24, 48, 72 hours after infusion, Cycle 1 Day 8, 15, 22:predose; Cycle 2 Day1: predose, 2, 6 h, 10, 24, 48, 72, 168 hours after infusion; Cycle 2 Day 15;Day 1 on Cycle 4, Cycle 6,Cycle 8: predose (each cycle is 28 days)
  The ratio of the drug exposure at a steady state to the drug exposure after the first administration.

SECONDARY OUTCOMES:
Adverse Events (AE) rate | From date of the first dose until the date of 30 days after last dose or new anti-tumor treatment, whichever came first
  The occurrence and severity of all AEs
Objective Response Rate (ORR) | Up to 2 years
  Defined as the percentage of Complete Response (CR) plus partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria
Duration of Response (DOR) | Up to 3 years
  Defined as the time from first documented response to documented disease progression.
Progression-free survival (PFS) | Up to 3 years
  Defined as the time from the first dose of TQB2922 to the first occurrence of disease progression or death from any cause.
Incidence of anti-drug antibody (ADA) | From the time of informed consent signed through 90 days after the last dose.
  Incidence of anti-drug antibody (ADA)

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China hospital, Sichuan University, Chengdu, Sichuan
  - Chengdu Third People's Hospital, Chengdu, Sichuan